CLINICAL TRIAL: NCT04076033
Title: Reliability, Reproducibility, and Efficiency of Functional Compressive Assessment in the Treatment of Secondary Lymphedema to the Treatment of Breast Cancer
Brief Title: Reliability and Reproducibility of Bandaging in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elaine Caldeira de Oliveira Guirro (Other)
Responsible Party: Sponsor-Investigator, Elaine Caldeira de Oliveira Guirro, Clinical professor, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 000001
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Functional Compressive Bandage; Lymphedema; Physiotherapy
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECF ESPIRAL (Experimental): The volunteer is submitted to four-layer spiral functional compressive bandage, then performs Taylor's Jebsen manual function test with comprehensive functional bandage (ECF).
  Interventions: Other: functional compressive bandage
- ECF OITO (Experimental): The volunteer is submitted to functional compressive bandage in eight with four layers, then performs the Taylor Jebsen manual function test with the comprehensive functional bandage (ECF).
  Interventions: Other: functional compressive bandage

INTERVENTIONS:
Other: functional compressive bandage — The functional compressive bandage is being performed with the volunteer sitting with the upper limb homolateral to the surgery supported by a support. After hydration of the limb, a cotton mesh is being used to prevent friction of the 1 cm density foam band being wrapped around the limb. No therapeutic procedure is being performed prior to functional compressive bandage.
  The bandage of the limb is being performed with 5 cm, 10 cm, 15 cm elastic cotton bandages from the fingers to the axillary region in four layers.

SUMMARY:
Functional Compressive Bandage (ECF) is a widely used therapeutic resource in the control of lymphedema resulting from the treatment of breast cancer, however, the effects inherent to the technique depend on the quality of the application. The aim of the study is to evaluate the reliability, reproducibility, and efficiency of treatment with different techniques in two studies. The first step aims to evaluate the reliability and reproducibility of the technique. The analysis of the pressure exerted by the four-layer bandage, applied by two evaluators previously trained and familiar with the ECF technique will perform the evaluations on the same volunteers in two moments, with an interval of one week between them. The intraclass correlation coefficient will be used to determine intra- and inter-examiner reliability, with its respective 95% confidence interval, standard error of measurement and minimum detectable change. The second stage aims to verify the efficiency of different ECF techniques in the functionality and circulation of the upper limb affected by lymphedema. This step is being performed by a single evaluator, and the ECF efficiency tested by the random application of two different techniques (spiral and eight), with a seven-day interval, and pressure assessment in mmHg. Upper limb functionality analysis is being performed using the Jebsen Taylor test performed before and with ECF on both limbs. The evaluation of the influence of the bandage in the circulation evaluated by Doppler ultrasound, before and after the test application. Member dominance assessed using the Edinburgh inventory.

DETAILED DESCRIPTION:
Functional Compressive Bandage (ECF) is a widely used therapeutic resource in the control of lymphedema resulting from the treatment of breast cancer, however, the effects inherent to the technique depend on the quality of the application. The aim of the study is to evaluate the reliability, reproducibility, and efficiency of treatment with different techniques in two studies. To this end, 50 volunteers will be evaluated, aged between 40 and 70 years, submitted to breast cancer treatment. The analyzes will be performed in two subprojects, conducted with randomized cross over design and seven days wash out period, so far 19 volunteers were collected. The first step aims to evaluate the reliability and reproducibility of the technique. The analysis of the pressure exerted by the four-layer bandage, applied by two evaluators previously trained and familiar with the ECF technique will perform the evaluations on the same volunteers in two moments, with an interval of one week between them. The intraclass correlation coefficient (ICC2,1) will be used to determine intra- and inter-examiner reliability, with its respective 95% confidence interval, standard measurement error and minimum detectable change. The second stage aims to verify the efficiency of different ECF techniques in the functionality and circulation of the upper limb affected by lymphedema. This step is being performed by a single evaluator, and the ECF efficiency tested by the random application of two different techniques (spiral and eight), with a seven-day interval, and pressure assessment in mmHg. Upper limb functionality analysis is being performed using the Jebsen Taylor test performed before and with ECF on both limbs. The evaluation of the influence of the bandage in the circulation evaluated by Doppler ultrasound, before and after the test application. Member dominance assessed using the Edinburgh inventory. Partial data was verified by descriptive analysis with mean and standard deviation. Data processing was performed using SPSS® software, version 13.0 (Chicago, IL, USA). A significance level of 5% was considered. The information obtained in the study aims to show the partial results of the preliminary and descriptive evaluation of the physical therapy intervention in women affected by lymphedema resulting from breast cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are age over 21 years, treatment for unilateral breast cancer, unilateral lymphedema resulting from treatment for breast cancer.

Exclusion Criteria:

* The exclusion criteria established are skin disorders; diabetes; adjuvant treatment in progress; submitted to bilateral axillary dissection; diagnosis of metastasis and at risk of peripheral arterial disease, functional change of upper limbs before breast cancer treatment.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 2 minutes
  mmHg

SECONDARY OUTCOMES:
Blood flow | 10 minutes
  mL/s
Jebsen Taylor test | 10 minutes
  time

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Caldeira de Oliveira Guirro, PhD, Study Director — University of Sao Paulo
Locations (1):
- University of São Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided